CLINICAL TRIAL: NCT06026527
Title: Intra-operative Magnesium Sulphate for Post-operative Pain in Patients Undergoing Total Abdominal Hysterectomy Under General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Priyanka Dahal, MD Resident- Anaesthesiology, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MagSulf1234
Record Dates: First submitted 2023-08-29; First posted 2023-09-07 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Post-operative Pain
Keywords: Magnesium, Pain, NRS, Abdominal hysterectomy, MgSO4
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Experimental): Magnesium group
  Interventions: Drug: Magnesium sulfate
- Group C (Placebo Comparator): Control group
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium sulfate — 50 mg/kg Magnesium sulphate in 93-95 ml Normal Saline ( making a total of 100 ml solution )will be infused intravenously over 20-30 minutes in the participants allocated to M group starting from the moment of induction of anaesthesia
  Other Names: Magnesium sulphate
  Arms: Group M
Drug: Normal Saline — 100 ml Normal Saline will be infused intravenously over 20-30 minutes in the participants allocated to control group starting from the moment of induction of anaesthesia
  Other Names: NS
  Arms: Group C

SUMMARY:
Post-operative pain management is a complex entity. It is one of the most critical parameters in the enhanced recovery after surgery protocol. Adequate postoperative pain relief leads to earlier mobilisation, shortened hospital stay, reduced hospital costs and increased patient satisfaction.

For post-operative analgesia, opioids have long been the mainstay of drugs used; however, they produce unwanted side effects, such as respiratory depression, nausea, vomiting and dependence. The major goal in postoperative pain management is to minimise the dose of a single medication and lessen its side effects, while still providing adequate analgesia by the use of multimodal analgesia. Paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), regional techniques like epidural analgesia, different kind of blocks and local wound infiltration are some of the components of multimodal approach to post- operative analgesia.

Besides, there are some drugs that may be used as adjuvants to opioids to enhance the analgesic efficacy and facilitate opioid sparing with a reduction in opioid related side effects. Magnesium sulphate, due to its N- Methyl D- Aspartate (NMDA) blocking property, has been studied as one of such non opioid adjuvants. The outcome of many of these studies is in favour of magnesium sulphate but there are negative reports as well.

So, in this study the investigators aim to evaluate the efficacy of intra-operative intravenous magnesium sulphate for post-operative pain and opioid use in patients undergoing abdominal hysterectomy under general anaesthesia.

DETAILED DESCRIPTION:
All women who have been planned for total abdominal hysterectomy will be enrolled in the study. Patients who do not meet the inclusion criteria or those who refuse to participate will be excluded from study . Other enrolled patients who meet the eligibility criteria will be randomised and allocated to two study groups- Magnesium (M) group and Control (C) group by computer generated numbers that will be concealed in a sequentially numbered, opaque sealed envelopes. The envelopes will be opened before the surgery begins by a doctor not involved in the study and not assigned to the Gynaecology operating room. The drug will be prepared and labelled study drug as: In group M- Magnesium sulphate @ 50mg/ kg in 100 ml of normal saline and in group C- 100 ml of normal saline. Anaesthetic management, administration of the study drug and any intra-operative changes in vitals requiring treatment will be recorded in the anaesthesia management sheet by another doctor who is assigned to Gynaecology operating room.

A day prior to surgery, eligible patients will be explained in detail about the purpose of study, need, benefits and risks of procedure. The participants will be explained about numerical rating scale (NRS) of pain, how to use it and rate it during post-operative period. Written informed consent will be obtained. The patients will be counselled about fasting protocol and asked to remain nil per oral of 2 hours for clear liquid, 6 hours for light foods and 8 hours for fatty food.

In pre-operative holding area : Baseline vitals systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP), heart rate (HR), respiratory rate (RR), Oxygen saturation (SpO2) will be recorded. Intravenous access will be established with an 18 or 20 gauge cannula. A 3-way stopcock will be attached to the cannula and Lactated Ringer's will be infused @ 100ml/hr.

In the operating room: Standard American Society of Anaesthesiologists monitors will be attached. All patients will be subjected to a standardised anaesthetic protocol. Induction of general anaesthesia, intubation, ventilation parameter set up and maintenance of anaesthesia will be done as per standard anaesthetic practice in our institute.

Meanwhile, at the time of induction, 100 ml of study drug will be infused via side port of 3-way stopcock over 20-30 minutes. Ringer lactate solution will be infused throughout the surgery as per standard practice in our institute. Hemodynamic parameters SBP, DBP, HR, SpO2, RR will be monitored and recorded as per anaesthesia protocol. Additional analgesia during the peri-operative period will be standardised with IV Paracetamol 15 mg/kg post induction and IV Fentanyl 0.5 mcg/kg every hour of intra-operative period and any additional dosing of analgesia will be recorded. Urine output monitoring will be done on hourly basis. If less than 0.5 ml/kg/hr, underlying cause will be looked for, and if no other causes is found, Mg toxicity will be suspected and serum magnesium level will be sent. Meanwhile necessary medical management will be done. Post operative nausea and vomiting (PONV) prophylaxis will be standardised in both groups of patient. IV Ondansetron 4mg single dose 15 to 20 minutes before extubation will be given. 0.25% Bupivacaine not exceeding 2 mg/kg dose will be administered locally at the site of surgical incision at the end of surgery. Reversal of muscle relaxation and extubation will be done as per attending anaesthesiologist. Patient will be transferred to recovery room.

Post operatively: Patients will be held in recovery room until adequate recovery from anaesthesia as judged by the Modified Aldrete Score. Score ≥ 9 will be deemed adequate. Post operative pain assessment will be done with Numerical Rating Scale (NRS). The NRS is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Pain assessment will be done by the attending nurse at time 0, 1, 6, 12, 18, 24 hours. The time 0 will be the first assessment of pain done in the recovery room once the patient is fully awake. If NRS > 3 at any time within 24 hours, IV Tramadol 50 mg will be given as rescue analgesia. NRS and vitals at this point will be recorded. If NRS > 3 even after 10 minutes of rescue analgesic , second dose of 50 mg of IV Tramadol up to a total dose of 150 mg including the initial bolus will be given.Vitals SBP, DBP, MAP, HR, RR, SpO2 will be monitored and recorded at 0, 1, 6, 12, 18, 24 hours. 24 hours total opioid consumption post-operatively will be recorded. Side effects of magnesium sulphate including nausea/ vomiting, flushing, hypotension, bradycardia, blurring of vision, decreased respiratory rate , muscle weakness, loss of deep tendon reflexes will be recorded and managed as per protocol.

Maintenance analgesia will be standardised as : IV Paracetamol 15 mg/kg every 6 hours and IV Ketorolac 30mg every 8 hours. For postoperative nausea and vomiting, IV Ondansetron 4 mg will be given every 8 hours as standard practice.

Management of the patients for any side effects will be done as described below:

Hypotension with SBP < 90 mmHg will be managed with IV Mephentermine 6mg bolus and repeated as required.

Bradycardia with HR < 50 beats/min will be managed with IV Atropine 0.6 mg bolus.

Respiratory depression will be graded as mild (RR 10-12), moderate (RR 8-10) and severe ( RR <8). Oxygen @ 6 L/ minute will supplemented via face mask. In case of severe respiratory depression, serum magnesium level will be sent in suspicion magnesium toxicity. If magnesium level comes out to be normal, respiratory depression due to opioid will be suspected and IV naloxone 0.4 mg will be given and repeated 2-3 minutes until RR rises above 8. Total naloxone dose will not exceed 10 mg.

Sedation will be quantified according to Pasero Opioid-induced Sedation Scale ( POSS) . In case of POSS >3, IV Naloxone will be infused as mentioned earlier.

If milder signs of hypermagnesemia like nausea, dizziness, confusion is noticed, it will be recorded and informed to the principal investigator. Meanwhile serum Magnesium level will be sent. The principal investigator will then attend the patient for signs of moderate hypermagnesemia and manage accordingly. Patients with normal renal function clinically assessed as urine output >0.5ml/kg/hour and mild hypermagnesemia will require no treatment. If signs of moderate hypermagnesemia occur, the principal investigator will attend the case for close monitoring of the ECG, blood pressure, neuromuscular function and respiratory function. If either hyporeflexia assessed as loss of patellar reflex, respiratory depression or changes in ECG is noticed individually or all at once, IV normal saline at 150 ml/hour and IV calcium gluconate 1 gm over 5 minutes will be infused. The rationale is that the actions of magnesium in neuromuscular and cardiac function become antagonized by calcium. In absence of improvement, same dose will be repeated. In case of severe hypermagnesemia, intravenous loop diuretic, IV Furosemide 1 mg/kg will be given to increase renal magnesium excretion.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective abdominal hysterectomy.
* Between the ages of 18- 65.
* American Society of Anesthesiologists Physical Status (ASA PS) I and II.

Exclusion Criteria:

* Neurological and psychiatric disorder.
* Drug or alcohol abuse.
* Patients with a known or suspected allergy to magnesium sulphate.
* Patients with any contraindication to magnesium sulphate (heart blocks, neuromuscular diseases)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of magnesium sulphate for post-operative pain | At 0, 1, 6,12 18 and 24 hours post-operatively
  Post operative pain will be assessed by using Numerical rating score (NRS) of pain. The NRS is a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Comparison of Numerical Rating Scale (NRS) score of pain | at 0, 1, 6, 12, 18, 24 hours post-operatively
  Comparison of Numerical Rating Scale score between Magnesium and control group.The NRS is a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Opioid as rescue analgesic use | The time to first rescue analgesic use within 24 hours post-operatively will be noted
  To compare the timing of first rescue analgesic used
Total opioid use | within 24 hours post-operatively
  Comparison of total opioid used between two groups
Side effects | within 24 hours post-operatively
  To determine any side effects of magnesium sulphate

CONTACTS AND LOCATIONS:
Overall Officials: Subhash P Acharya, MD FACC FCCP, Study Chair — Tribhuvan University Teaching Hospital; Bashu D Parajuli, MD, FOA, Study Chair — Tribhuvan University Teaching Hospital; Pankaj Joshi, MD, FLTA (ICA), Study Chair — Tribhuvan University Teaching Hospital; Priyanka Dahal, MD Resident, Principal Investigator — Tribhuvan University Teaching Hospital
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shekhar C, Paswan B, Singh A. Prevalence, sociodemographic determinants and self-reported reasons for hysterectomy in India. Reprod Health. 2019 Aug 2;16(1):118. doi: 10.1186/s12978-019-0780-z. PMID 31375139
- [Background] Clarke-Pearson DL, Geller EJ. Complications of hysterectomy. Obstet Gynecol. 2013 Mar;121(3):654-673. doi: 10.1097/AOG.0b013e3182841594. PMID 23635631
- [Background] Perniola A, Gupta A, Crafoord K, Darvish B, Magnuson A, Axelsson K. Intraabdominal local anaesthetics for postoperative pain relief following abdominal hysterectomy: a randomized, double-blind, dose-finding study. Eur J Anaesthesiol. 2009 May;26(5):421-9. doi: 10.1097/EJA.0b013e3283261b53. PMID 19521298
- [Background] Chung F, Ritchie E, Su J. Postoperative pain in ambulatory surgery. Anesth Analg. 1997 Oct;85(4):808-16. doi: 10.1097/00000539-199710000-00017. PMID 9322460
- [Background] Kehlet H, Dahl JB. The value of "multimodal" or "balanced analgesia" in postoperative pain treatment. Anesth Analg. 1993 Nov;77(5):1048-56. doi: 10.1213/00000539-199311000-00030. No abstract available. PMID 8105724
- [Background] White PF. The role of non-opioid analgesic techniques in the management of pain after ambulatory surgery. Anesth Analg. 2002 Mar;94(3):577-85. doi: 10.1097/00000539-200203000-00019. No abstract available. PMID 11867379
- [Background] Woolf CJ, Thompson SWN. The induction and maintenance of central sensitization is dependent on N-methyl-D-aspartic acid receptor activation; implications for the treatment of post-injury pain hypersensitivity states. Pain. 1991 Mar;44(3):293-299. doi: 10.1016/0304-3959(91)90100-C. PMID 1828878
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Background] Tramer MR, Schneider J, Marti RA, Rifat K. Role of magnesium sulfate in postoperative analgesia. Anesthesiology. 1996 Feb;84(2):340-7. doi: 10.1097/00000542-199602000-00011. PMID 8602664
- [Background] Wilder-Smith CH, Knopfli R, Wilder-Smith OH. Perioperative magnesium infusion and postoperative pain. Acta Anaesthesiol Scand. 1997 Sep;41(8):1023-7. doi: 10.1111/j.1399-6576.1997.tb04830.x. PMID 9311401
- [Background] Ko SH, Lim HR, Kim DC, Han YJ, Choe H, Song HS. Magnesium sulfate does not reduce postoperative analgesic requirements. Anesthesiology. 2001 Sep;95(3):640-6. doi: 10.1097/00000542-200109000-00016. PMID 11575536
- [Background] Kara H, Sahin N, Ulusan V, Aydogdu T. Magnesium infusion reduces perioperative pain. Eur J Anaesthesiol. 2002 Jan;19(1):52-6. doi: 10.1017/s026502150200008x. PMID 11913804
- [Background] Feld JM, Laurito CE, Beckerman M, Vincent J, Hoffman WE. Non-opioid analgesia improves pain relief and decreases sedation after gastric bypass surgery. Can J Anaesth. 2003 Apr;50(4):336-41. doi: 10.1007/BF03021029. English, French. PMID 12670809
- [Background] Taheri A, Haryalchi K, Mansour Ghanaie M, Habibi Arejan N. Effect of low-dose (single-dose) magnesium sulfate on postoperative analgesia in hysterectomy patients receiving balanced general anesthesia. Anesthesiol Res Pract. 2015;2015:306145. doi: 10.1155/2015/306145. Epub 2015 Feb 1. PMID 25705223
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Hammond DA, Stojakovic J, Kathe N, Tran J, Clem OA, Erbach K, King J. Effectiveness and Safety of Magnesium Replacement in Critically Ill Patients Admitted to the Medical Intensive Care Unit in an Academic Medical Center: A Retrospective, Cohort Study. J Intensive Care Med. 2019 Nov-Dec;34(11-12):967-972. doi: 10.1177/0885066617720631. Epub 2017 Jul 13. PMID 28703019
- [Background] Yamaguchi H, Shimada H, Yoshita K, Tsubata Y, Ikarashi K, Morioka T, Saito N, Sakai S, Narita I. Severe hypermagnesemia induced by magnesium oxide ingestion: a case series. CEN Case Rep. 2019 Feb;8(1):31-37. doi: 10.1007/s13730-018-0359-5. Epub 2018 Aug 22. PMID 30136128
- [Background] Kobelt P, Burke K, Renker P. Evaluation of a standardized sedation assessment for opioid administration in the post anesthesia care unit. Pain Manag Nurs. 2014 Sep;15(3):672-81. doi: 10.1016/j.pmn.2013.11.002. Epub 2014 Jan 22. PMID 24461253
- [Background] BELLVILLE JW, BROSS ID, HOWLAND WS. A method for the clinical evaluation of antiemetic agents. Anesthesiology. 1959 Nov-Dec;20:753-60. doi: 10.1097/00000542-195911000-00002. No abstract available. PMID 13798617
- [Background] Blaine J, Chonchol M, Levi M. Renal control of calcium, phosphate, and magnesium homeostasis. Clin J Am Soc Nephrol. 2015 Jul 7;10(7):1257-72. doi: 10.2215/CJN.09750913. Epub 2014 Oct 6. PMID 25287933